CLINICAL TRIAL: NCT03016585
Title: Effectiveness of Tai Chi on Cardiac Autonomic Function and Symptomatology in Women With Fibromyalgia: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Collaborators: Marymount University (Other)
Responsible Party: Principal Investigator, Won-mok son, Ph.D, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PusanNU
Record Dates: First submitted 2017-01-08; First posted 2017-01-10 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

ARMS (2):
- Tai Chi Training (Experimental): Tai Chi exercises 3 times per wk for 12 weeks
  Interventions: Other: Tai Chi Training
- Control (No Intervention): This arm involves not making any change to the subject's lifestyle at the moment of the start of the intervention and for 12 weeks.

INTERVENTIONS:
Other: Tai Chi Training — Participants practiced, under supervised instruction, 10 forms from the classic Yang style of Tai Chi 3 times per wk for 12 weeks.The Tai Chi sessions lasted approximately 55 minutes and included a 10-minute warm up, 40 minutes of practice and exercise finalizing with a 5-minute cooldown period.
  Arms: Tai Chi Training

SUMMARY:
Fibromyalgia (FM) is an idiopathic disease affecting approximately 3% of the world population, primarily diagnosed in middle-aged women. Although FM is mainly characterized by chronic pain and fatigue, reduced muscular strength and flexibility are common symptoms associated with the presentation of the disorder. Interestingly, the etiology and underlying mechanism of FM are not completely understood, but previous findings suggest that autonomic dysfunction may explain some of the FM symptoms.

Compared to age-matched healthy individuals, patients with FM have an attenuated autonomic function which is associated with a reduction in vagal tone and increase in sympathetic activity. Therefore, autonomic function is a worthwhile target intervention in individuals with FM. Although traditional exercise ( both aerobic and resistance) has been shown to effectively improve HRV parameters and FM symptoms, most FM patients display a decline in adherence to traditional exercise and continue to experience considerable pain and fatigue years after the original diagnosis ultimately requiring medication to control their symptoms.Thus, new approaches are needed to improve autonomic function and clinical symptoms in patients with FM, which will ultimately improve their physical and emotional functioning leading to a better quality of life.

Tai Chi (TC) is a form of ancient Chinese martial art which integrates slow movements, controlled breathing and mental concentration. TC training is safe for special populations and has previously shown to decrease pain, fatigue as well as other FM related symptoms.However, the potential role of TC training on autonomic function is largely unexplored.

The investigators hypothesis is that 12 weeks of TC training would improve our primary outcome of autonomic function through improvements in sympathovagal balance, and the secondary outcomes measures of FM symptoms (pain, fatigue and sleep quality), strength and flexibility.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of 12 weeks of TC training on on cardiac autonomic function, FM symptoms (pain, fatigue and sleep quality), strength and flexibility. The specific aim of the study is:

- To evaluate the effects of 12 weeks of TC training on autonomic function arterial function by assessing heart rate variability

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia
* Sedentary

Exclusion Criteria:

* Known pulmonary, cardiovascular, renal, adrenal, pituitary, severe psychiatric or thyroid diseases.
* Use of hormone replacement therapy during the 6 months prior to the study.
* Any medication changes in the previous 12 months.
* Current participation in psychological or physical therapy
* History of steady exercise or received exercise training in the last year

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Autonomic Function | 12 weeks
  Heart Rate Variability was assessed from electrocardiogram

SECONDARY OUTCOMES:
Fibromyalgia Symptomatology | 12 weeks
  Subjects filled visual analog scales (VAS) to evaluate symptom severity before and after 12 weeks.
Flexibilty | 12 weeks
  Flexibility was measured using the Sit and Reach Test
Muscle Strength | 12 weeks
  one repetition maximum (1RM) was performed using a leg extension machine